CLINICAL TRIAL: NCT01230593
Title: A 5-year Multicenter Prospective Randomized Trial Comparing Three Conservative Chalazion Treatments
Brief Title: Chalazion Conservative Treatment Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Edward-Elmhurst Health System (Other)
Responsible Party: Principal Investigator, Albert Wu, M.D. Ph.D., McMaster University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-469
Record Dates: First submitted 2010-10-27; First posted 2010-10-29 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Chalazion Unspecified Eye, Unspecified Eyelid; Chalazion Left Eye, Unspecified Eyelid; Chalazion Right Eye, Unspecified Eyelid; Chalazion Both Eyes
MeSH Terms: interventions — Ointments; Tobramycin; Tobramycin, Dexamethasone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hot Compress (Active Comparator): "Hot Compress"
  Interventions: Other: Hot Compresses
- Tobrex (Active Comparator): "Hot Compress", "Tobrex Drops", "Tobrex Ointment"
  Interventions: Drug: Hot Compress plus Tobramycin Drops and Ointment
- Tobradex (Active Comparator): "Hot Compress", "Tobradex Drops", "Tobradex Ointment"
  Interventions: Drug: Hot compress plus Tobramycin/Dexamethasone Drops and Ointment

INTERVENTIONS:
Drug: Hot Compress plus Tobramycin Drops and Ointment — In addition to hot compress, Tobramycin drops will be given to the affected eye 3x/day, and Tobramycin ointment will be given at night before bed.
  Other Names: Aktob; Tobralcon; Tobrasol; Tobramycin
  Arms: Tobrex
Drug: Hot compress plus Tobramycin/Dexamethasone Drops and Ointment — In addition to hot compress, Tobramycin/Dexamethasone drops will be given to the affected eye 3x/day, and Tobramycin/Dexamethasone ointment will be given at night before bed.
  Other Names: Tobramycin/dexamethasone
  Arms: Tobradex
Other: Hot Compresses — Hot compresses 3x/day to eyelids
  Arms: Hot Compress

SUMMARY:
An eyelid stye, or chalazion, is the most common eyelid ailment, and is caused by the blockage of one of the oil secreting glands of the eyelid (meibomian glands). This leads to a typically painful, swollen, and red eyelid bump that lasts from days to weeks and months. The chalazion may cause tearing, pressure on the cornea, and irritation, all of which contribute to its morbidity. There are many anecdotal first line treatments for this condition, including warm compresses to the eyelid, topical antibiotics, topical steroids, topical combination antibiotic/steroid, and oral antibiotics. There have been no clinical trials to compare the efficacy of any of these conservative treatments. We wish to determine the most effective conservative medical treatment for chalazia.

ELIGIBILITY:
Inclusion Criteria

* Patients age 18 and above
* Patient with a palpable chalazion on any eyelid
* Patients with multiple chalazia but only a single one on each lid
* Normal lid anatomy enabling lid eversion

Exclusion Criteria

* Patients with chalazia with atypical features (recurring chalazion, abnormal surrounding lid tissue, associated loss of lashes) that may indicate suspicion of malignancy
* Patients allergic to any agents being used in the study (tobramycin, dexamethasone)
* Patients who have had previous eyelid surgery to the same eyelid as the chalazion
* Patients under 18 years of age
* Patients without palpable lid chalazion
* Patients with multiple chalazia on one eyelid
* Patients with concurrent eyelid infection (cellulitis or conjunctivitis)
* Patients unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-11; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Y Wu, M.D., Ph.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (2):
  - Elmhurst Hospital Center, Elmhurst, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
- St. Joseph's Hospital Eye Clinic, Stoney Creek, Ontario, Canada

REFERENCES:
- [Derived] Wu AY, Gervasio KA, Gergoudis KN, Wei C, Oestreicher JH, Harvey JT. Conservative therapy for chalazia: is it really effective? Acta Ophthalmol. 2018 Jun;96(4):e503-e509. doi: 10.1111/aos.13675. Epub 2018 Jan 16. PMID 29338124

RESULTS

PARTICIPANT FLOW:
Groups:
- Hot Compress: Patients in the hot compress arm will be shown how to apply hot compresses to the affected lid and gently massage the lid to encourage the chalazion to spontaneously drain for 5 minutes, 3x/day.
  Hot Compresses: Hot compresses 3x/day to eyelids
- Hot Compress + Tobramycin Drops and Ointment: In addition to using hot compress, patients in the Tobramycin arm will be prescribed Tobramycin drops 3x/day and ointment to be applied before bedtime.
  Tobramycin Drops and Ointment: Tobramycin drops will be given to the affected eye 3x/day, and Tobramycin ointment will be given at night before bed.
- Hot Compress + Tobramycin/Dexamethasone Drops and Ointment: In addition to using hot compress, patients in the Tobramycin/Dexamethasone arm will be prescribed Tobramycin/Dexamethasone drops 3x/day and ointment to be applied before bedtime.
  Tobramycin/Dexamethasone Drops and Ointment: Tobramycin/Dexamethasone drops will be given to the affected eye 3x/day, and Tobramycin/Dexamethasone ointment will be given at night before bed.
Period: Overall Study
Arm/Group | Hot Compress | Hot Compress + Tobramycin Drops and Ointment | Hot Compress + Tobramycin/Dexamethasone Drops and Ointment
Started | 50 | 50 | 50
Completed | 35 | 32 | 38
Not Completed | 15 | 18 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hot Compress | Hot Compress + Tobramycin Drops and Ointment | Hot Compress + Tobramycin/Dexamethasone Drops and Ointment | Total
Number analyzed (Participants) | 50 | 50 | 49 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.50 (15) | 46.42 (19) | 47.52 (17) | 47.41 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 30 | 79
  Male | 25 | 26 | 19 | 70
Region of Enrollment [Number; unit: participants]
  Canada | 8 | 5 | 14 | 27
  United States | 42 | 45 | 35 | 122
Pre-treatment lesion duration (months) [Mean (Standard Deviation); unit: months] | 3.55 (6) | 2.88 (3) | 5.72 (13) | 3.96 (8)
Initial lesion size (mm) [Mean (Standard Deviation); unit: millimeters] | 6.05 (3) | 6.16 (3) | 6.38 (3) | 6.19 (3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Resolution
Description: Defined as number of patients with chalazion size regression of 100%
Time Frame: 4-6 weeks
Population: Intention to treat population
Measure: Number; unit: participants
Arm/Group | Hot Compress | Hot Compress + Tobramycin Drops and Ointment | Hot Compress + Tobramycin/Dexamethasone Drops and Ointment
Number analyzed (Participants) | 50 | 50 | 49
participants | 13 | 12 | 11

2. Secondary Outcome: Chalazion Size Difference Post-Treatment
Description: Change of size of eyelid chalazion in millimeters from baseline to 4-6 weeks post-treatment
Time Frame: baseline and 4-6 weeks
Population: Intention to treat population
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Hot Compress | Hot Compress + Tobramycin Drops and Ointment | Hot Compress + Tobramycin/Dexamethasone Drops and Ointment
Number analyzed (Participants) | 50 | 50 | 49
millimeters | 1.20 (3) | 1.69 (3) | 1.54 (3)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored over a time frame of 4-6 weeks from baseline enrollment of each participant. Participants returned for follow-up between 4 and 6 weeks after starting treatment.
Description: Serious Adverse Events
Groups:
- Hot Compress, Tobrex Drops, Tobrex Ointment: In addition to using hot compress, patients in the Tobramycin arm will be prescribed Tobramycin drops 3x/day and ointment to be applied before bedtime.
  Tobramycin Drops and Ointment: Tobramycin drops will be given to the affected eye 3x/day, and Tobramycin ointment will be given at night before bed.
- Hot Compress, Tobradex Drops, Tobradex Ointment: In addition to using hot compress, patients in the Tobramycin/Dexamethasone arm will be prescribed Tobramycin/Dexamethasone drops 3x/day and ointment to be applied before bedtime.
  Tobramycin/Dexamethasone Drops and Ointment: Tobramycin/Dexamethasone drops will be given to the affected eye 3x/day, and Tobramycin/Dexamethasone ointment will be given at night before bed.
Arm/Group | Hot Compress | Hot Compress, Tobrex Drops, Tobrex Ointment | Hot Compress, Tobradex Drops, Tobradex Ointment
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
Large loss to follow-up - only 70% completed follow-up - was a limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No